CLINICAL TRIAL: NCT00330135
Title: Multicentre, Randomized, Placebo-Controlled, Double-Blind Clinical Trial to Investigate the Efficacy of Sodium Hyaluronate in Patients With Symptomatic Hip Osteoarthritis
Brief Title: The Efficacy Study of Sodium Hyaluronate to Treat Symptomatic Hip Osteoarthritis
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Catherine Koch, Daiichi Sankyo France
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ADA 2003-01
Record Dates: First submitted 2006-05-23; First posted 2006-05-25 (Estimated); Last update posted 2008-01-09 (Estimated); Status verified 2008-01

CONDITIONS: Symptomatic Hip Osteoarthritis
Keywords: hip osteoarthritis; Hyaluronic acid; Viscosupplementation; intra-articular injections
MeSH Terms: conditions — Osteoarthritis, Hip | interventions — Hyaluronic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Sodium hyaluronate 2.5 ml - 1 injection
  Interventions: Drug: Sodium hyaluronate
- 2 (Placebo Comparator): Placebo injection - 1 injection
  Interventions: Drug: placebo injection

INTERVENTIONS:
Drug: Sodium hyaluronate — Sodium hyaluronate 2.5 ml - 1 injection
  Arms: 1
Drug: placebo injection — placebo injection - 1 injection
  Arms: 2

SUMMARY:
To demonstrate the difference in terms of symptomatic efficacy between ADANT® sodium hyaluronate and placebo following an intra-articular injection in patients with symptomatic osteoarthritis of the hip.

Each patient will receive an injection of sodium hyaluronate or placebo in the symptomatic hip and will be followed up for three months.

At the third month, if the score for overall pain is still > 40 mm on the VAS, a second injection of ADANT® can be given irrespective of which treatment was received previously. The patient will be followed up for a further 3 months in an open-label fashion (monthly visits).

ELIGIBILITY:
Inclusion Criteria:

* 1. Primary osteoarthritis of the hip defined according to the ACR criteria; symptomatic, 2. Osteoarthritis of radiological grade II to III according to the Kellgren-Lawrence classification, using X-rays performed during the last three months, 3. Overall pain intensity between 40 and 80 mm on a VAS of 100 mm at the pre-screening examination, 4. The patients experienced pain at least one in two days during the last 30 days, it was resistant to paracetamol treatment at a dose of 4 g/day and a step 2 analgesic or a NSAID taken for at least 10 days, 5. A prosthesis is not planned in the next six months.

Exclusion Criteria:

* Women who are pregnant or breastfeeding or women who could become pregnant and are not using effective contraception,
* Major dysplasia (defined using Lequesne's criteria as dislocation of the hip),
* Treatment by intra-articular injection of hyaluronic acid in the symptomatic hip during the 6 months prior to pre-screening,
* Patients with a history of hypersensitivity to any of the ingredients in the hyaluronan,
* The presence of inflammatory arthropathy or another disorder or condition that could affect the joint (e.g., rheumatoid arthritis, metabolic bone disease, femoral head necrosis, psoriasis, gout, infection),
* Another muscular or skeletal condition that could interfere with the evaluation of the efficacy of the treatment on the hip in question (evaluation of pain or functional handicap),
* Systemic corticosteroid therapy or intra-articular injection of corticosteroids into the ipsilateral hip or knee within the last month,
* Intermittent claudication or vascular disease,
* Previous surgery on the hip in question,
* Septic arthritis at any site,
* Any surgical procedure, including arthroplasty or arthroscopy, to the hip during the six months prior to pre-screening or surgery scheduled during the trial,
* Any chronic skin condition that could affect the site of the injection,
* Use of the investigational treatment or material during the last three months,
* Oral or injectable anticoagulant treatment,
* Antiaggregant platelet treatment, particularly low-dose aspirin,
* Symptomatic chondrocalcinosis in the painful hip

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2005-01; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Change in overall pain, 3 months after a single intra-articular injection. The intensity of the pain will be evaluated using a continuous VAS of 100 mm of the overall level of pain in the affected hip. | 3 months

SECONDARY OUTCOMES:
Proportion of responding patients and proportion of patients with a symptomatic response (OARSI criterion) | 3 months
WOMAC index (the 3 subscales) | 3 months
Consumption of analgesics and NSAIDs | 3 months
Evaluation of tolerability (AE reporting) | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Xavier Chevalier, Professor, Principal Investigator — Head of the department of rheumatology Hopital Henri Mondor, Creteil, France
Locations (1):
- Rueil-Malmaison, France

REFERENCES:
- [Derived] Richette P, Ravaud P, Conrozier T, Euller-Ziegler L, Mazieres B, Maugars Y, Mulleman D, Clerson P, Chevalier X. Effect of hyaluronic acid in symptomatic hip osteoarthritis: a multicenter, randomized, placebo-controlled trial. Arthritis Rheum. 2009 Mar;60(3):824-30. doi: 10.1002/art.24301. PMID 19248105